CLINICAL TRIAL: NCT04818385
Title: Prospective Observational Cohort Study of Patients With Moderate to Severe Chronic Plaque Psoriasis in Taiwan
Brief Title: Study to Assess the Change in Disease State When Subcutaneous Risankizumab Injection is Given to Adult Participants With Psoriasis in Taiwan
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P20-272
Record Dates: First submitted 2021-03-24; First posted 2021-03-26 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Psoriasis
Keywords: Psoriasis; Risankizumab; Skyrizi; Plaque Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Participants Receiving Risankizumab: Participants will receive risankizumab as prescribed by their physician.
- Participants Receiving All Other Biologics: Participants will receive all other biologics as prescribed by their physician.

SUMMARY:
Psoriasis (PsO) is a chronic, disease characterized by marked inflammation of the skin that results in thick, red, scaly plaques and is associated with high burden of illness that results in a negative impact on long-term health outcomes including quality of life (QoL). The main objective of this study is to characterize the durability of response of risankizumab compared to other biologics measured by the Psoriasis Area and Severity Index (PASI) 90 response in adult participants with moderate to severe chronic plaque psoriasis who are either new or have used a biological treatment in the past.

Risankizumab is a drug approved for the treatment of moderate-to-severe plaque psoriasis. Participants who are prescribed risankizumab or other comparator drugs in the real world setting are enrolled in this study. Data from a total of approximately 240 participants; 160 using risankizumab and 80 using other biologics will be evaluated across Taiwan.

Participants will receive subcutaneous risankizumab injection or or other biologic as prescribed by their physician. Data from these participants will be collected for approximately 2 years.

There may be a higher burden for participants in this study compared to standard of care. Participants will attend regular visits per routine clinical practice. The effect of the treatment will be checked by medical assessments, checking for side effects, and by questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of moderate to severe chronic plaque-type psoriasis diagnosed by a specialist t at the time of recruitment.
* Initiating an approved biologic treatment for psoriasis as per regulatory and reimbursement policy in Taiwan. Physician's decision with any of the above-mentioned treatments must have been reached prior to and independently of recruitment in the study.
* Treatments prescribed in accordance to both the product monograph, regulatory and reimbursement policies in Taiwan.

Exclusion Criteria:

- Participation in an interventional clinical trial, concurrently or within the last 30 days. Participation in another PMOS or Registry is acceptable.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with moderate to severe plaque psoriasis.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2021-05-31 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
The Percentage of Participants who Achieved Psoriasis Area and Severity Index (PASI) 90 | Week 24
  The PASI is defined based on the percent reduction from baseline, generally summarized as a dichotomous outcome based on achieving over an 90% reduction. The PASI is used to evaluate a participant's overall psoriasis disease state that includes the percent of surface area of skin that is affected and the severity of erythema, infiltration, and desquamation over four body regions (head, upper extremities, trunk, and lower extremities). Scores range from 0 to 72, with the highest score representing complete erythroderma of the severest degree.

SECONDARY OUTCOMES:
Time of First Treatment Change | Up to Week 108
  Time of first treatment change is defined as any treatment change including discontinuation, dose escalation and dosing interval shortening.
The Percentage of Participants who Achieved PASI 75 | Up to Week 108
  The PASI is defined based on the percent reduction from baseline, generally summarized as a dichotomous outcome based on achieving over an 75% reduction. The PASI is used to evaluate a participant's overall psoriasis disease state that includes the percent of surface area of skin that is affected and the severity of erythema, infiltration, and desquamation over four body regions (head, upper extremities, trunk, and lower extremities). Scores range from 0 to 72, with the highest score representing complete erythroderma of the severest degree.
The Percentage of Participants who Achieved PASI 90 | Up to Week 108
  The PASI is defined based on the percent reduction from baseline, generally summarized as a dichotomous outcome based on achieving over an 90% reduction. The PASI is used to evaluate a participant's overall psoriasis disease state that includes the percent of surface area of skin that is affected and the severity of erythema, infiltration, and desquamation over four body regions (head, upper extremities, trunk, and lower extremities). Scores range from 0 to 72, with the highest score representing complete erythroderma of the severest degree.
The Percentage of Participants who Achieved PASI 100 | Up to Week 108
  The PASI is defined based on the percent reduction from baseline, generally summarized as a dichotomous outcome based on achieving over an 100% reduction. The PASI is used to evaluate a participant's overall psoriasis disease state that includes the percent of surface area of skin that is affected and the severity of erythema, infiltration, and desquamation over four body regions (head, upper extremities, trunk, and lower extremities). Scores range from 0 to 72, with the highest score representing complete erythroderma of the severest degree.
Percentage of Participants who Achieved Absolute PASI<=5 | Up to Week 108
  The absolute PASI is used to assess the benefit of psoriasis therapy, with a higher score indicating a greater percent reduction.
Percentage of Participants who Achieved Absolute PASI<=3 | Up to Week 108
  The absolute PASI is used to assess the benefit of psoriasis therapy, with a higher score indicating a greater percent reduction.
Percentage of Participants who Achieved Absolute PASI<=1 | Up to Week 108
  The absolute PASI is used to assess the benefit of psoriasis therapy, with a higher score indicating a greater percent reduction.
The Percentage of Participants who Achieved Dermatology Life Quality Index (DLQI) 0/1 | Up to Week 108
  DLQI total score is calculated by summing the scores of each question resulting in a range of 0 to 30 where the higher the score, the more the quality of life is impaired.
Time to Achieved PASI 75 | Up to Week 108
  The PASI is defined based on the percent reduction from baseline, generally summarized as a dichotomous outcome based on achieving over an 75% reduction. The PASI is used to evaluate a participant's overall psoriasis disease state that includes the percent of surface area of skin that is affected and the severity of erythema, infiltration, and desquamation over four body regions (head, upper extremities, trunk, and lower extremities). Scores range from 0 to 72, with the highest score representing complete erythroderma of the severest degree.
Time to Achieved PASI 100 | Up to Week 108
  The PASI is defined based on the percent reduction from baseline, generally summarized as a dichotomous outcome based on achieving over an 100% reduction. The PASI is used to evaluate a participant's overall psoriasis disease state that includes the percent of surface area of skin that is affected and the severity of erythema, infiltration, and desquamation over four body regions (head, upper extremities, trunk, and lower extremities). Scores range from 0 to 72, with the highest score representing complete erythroderma of the severest degree.
Time to Achieved PASI 90 | Up to Week 108
  The PASI is defined based on the percent reduction from baseline, generally summarized as a dichotomous outcome based on achieving over an 90% reduction. The PASI is used to evaluate a participant's overall psoriasis disease state that includes the percent of surface area of skin that is affected and the severity of erythema, infiltration, and desquamation over four body regions (head, upper extremities, trunk, and lower extremities). Scores range from 0 to 72, with the highest score representing complete erythroderma of the severest degree.
The Percentage of Participants who Achieved PASI 90 at 24 Weeks and Maintained the Response Without Changing the Indicated Dose or Dosing Interval | Up to Week 108
  The PASI is defined based on the percent reduction from baseline, generally summarized as a dichotomous outcome based on achieving over an 90% reduction. The PASI is used to evaluate a participant's overall psoriasis disease state that includes the percent of surface area of skin that is affected and the severity of erythema, infiltration, and desquamation over four body regions (head, upper extremities, trunk, and lower extremities). Scores range from 0 to 72, with the highest score representing complete erythroderma of the severest degree.
Change from Baseline in PASI | Up to Week 108
  The PASI is used to evaluate a participant's overall psoriasis disease state that includes the percent of surface area of skin that is affected and the severity of erythema, infiltration, and desquamation over four body regions (head, upper extremities, trunk, and lower extremities). Scores range from 0 to 72, with the highest score representing complete erythroderma of the severest degree.
Change from Baseline in Body Surface Area (BSA) Affected by Psoriasis | Up to Week 108
  BSA affected by psoriasis as assessed by the Investigator.
Change from Baseline in DLQI | Up to Week 108
  DLQI total score is calculated by summing the scores of each question resulting in a range of 0 to 30 where the higher the score, the more the quality of life is impaired.
Number of Participants with Adverse Events (AE) | Up to Week 108
  An AE is defined as any untoward medical occurrence in a participant, which does not necessarily have a causal relationship with their treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not the event is considered causally related to the use of the product.
Time to Reach Absolute PASI 10 After Withdraw from Latest Biologic Therapy | Up to 5 years Medical Chart Review Prior to Enrollment
  The absolute PASI is used to assess the benefit of psoriasis therapy, with a higher score indicating a greater percent reduction.
Time to Reach Loss of PASI 50 After Withdraw from Latest Biologic Therapy | Up to 5 years Medical Chart Review Prior to Enrollment
  The PASI is defined based on the percent reduction from baseline, generally summarized as a dichotomous outcome based on achieving over an 50% reduction. The PASI is used to evaluate a participant's overall psoriasis disease state that includes the percent of surface area of skin that is affected and the severity of erythema, infiltration, and desquamation over four body regions (head, upper extremities, trunk, and lower extremities). Scores range from 0 to 72, with the highest score representing complete erythroderma of the severest degree.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (8):
- Taiwan (8):
  - National Taiwan University Hospital /ID# 230017, Taipei City, Taipei
  - National Taiwan University Hospital - Hsinchu branch /ID# 238432, Hsinchu
  - Hualien Tzu Chi Hospital /ID# 238431, Hualien City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital /ID# 230016, Kaohsiung City
  - China Medical University Hospital /ID# 229961, Taichung
  - National Cheng Kung University Hospital /ID# 253776, Tainan
  - Taipei Medical University Hospital /ID# 230018, Taipei
  - Linkou Chang Gung Memorial Hospital /ID# 253775, Taoyuan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.rxabbvie.com/